CLINICAL TRIAL: NCT04078451
Title: The Clinical Study of Laparoscopic Cholecystectomy With the Preservation of the Main Cystic Artery
Brief Title: Study of Left Side of Laparoscopic Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Luhe Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-LHKY-001-02
Record Dates: First submitted 2018-11-18; First posted 2019-09-06 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Cholecystitis
Keywords: cholecystectomy; Laparoscopic
MeSH Terms: conditions — Cholecystitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the experimental group (Experimental): The experimental group operated by the left side of laparoscopic cholecystectomy preserving the main cystic artery.
  The operation area of cystic artery dissection is moved from the traditional triangular area to the gallbladder neck plane, away from the hepatic duct and hepatic portal.Only the superficial and even more minute branches of the cystic artery were isolated and coagulated.
  Interventions: Procedure: preserve the main cystic artery
- the control group (No Intervention): treated with conventional laparoscopic cholecystectomy cutting the cystic artery

INTERVENTIONS:
Procedure: preserve the main cystic artery — The experimental group preserve the main cystic artery, and the control group cut off the main cystic artery
  Arms: the experimental group

SUMMARY:
Prospectively selected 100 cases of patients who suffered from gallstones ro cholecystic polypus and treated with laparoscopic cholecystectomy in our hospital. Randomly divided into the experimental group and the control group. The experimental group preserve the main cystic artery, and the control group treated with conventional laparoscopic cholecystectomy. Collection of statistics: including general data(gender, age, BMI, etc.), time of surgery, intraoperative blood loss, incidence of surgical complications (delayed hemorrhage, biliary injury, etc.) and postoperative pain score, etc.

DETAILED DESCRIPTION:
1. research object (1)patients who suffered from gallstones ro cholecystic polypus. (2)Informed and consented to participate in this clinical trial (3)Number of enrolled cases：100.（About 700 cases were treated in our hospital）
2. Inclusion criteria

(1) consistent with the indications of cholecystectomy (2) no cholangitis or pancreatitis (3) no diabetes (4) the operation time is less than or equal to 1 hour 3.Exclusion criteria

1. patients with acute cholecystitis
2. cystic arterial variation causes related complications
3. patients receiving analgesic drugs after surgery 4.research methods 4.1 Grouping method: random number table method was applied to randomly divide into 2 groups.

4.2 surgical method：Laparoscopic cholecystectomy with the preservation of the main cystic artery

1. General anesthesia, use laryngeal mask
2. making CO2 pneumoperitoneum through the superior border of umbilical pneumoperitoneum pressure 12 -- 14 mmHg(1 mmHg=0.(133 kPa), the puncture sleeve was placed under laparoscopy according to the three-hole method.
3. To expose the gallbladder triangle, cut the serous membrane of the triangular region along the gallbladder tube, expose the neck and the left half of the gallbladder tube, push the rest tissue of the triangular region (including the main cystic artery, etc.) to the right, and separate the right half of the gallbladder tube, exposing the whole gallbladder tube.
4. Cutting off after clipping the gallbladder tube;
5. Turn up the gallbladder neck, cut off the superficial and deep branches of the gallbladder artery by electric hook along the gallbladder wall.
6. Remove the gallbladder. through the umbilical hole and close the puncture hole. 4.3 main outcome measures

(1) General data of patients (gender, age, BMI, etc.); (2) Operation time, intraoperative blood loss, surgical complications (delayed hemorrhage, biliary tract injury, etc.) incidence.

ELIGIBILITY:
Inclusion Criteria:

1. consistent with the indications of cholecystectomy
2. no cholangitis or pancreatitis
3. no diabetes
4. the operation time is less than or equal to 1 hour

Exclusion Criteria:

1. patients with acute cholecystitis
2. cystic arterial variation causes related complications
3. patients receiving analgesic drugs after surgery

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-30 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Operation time | One hour to 24 hours after surgery
  Compare the operation time between the two operations
intraoperative blood loss | One hour to 24 hours after surgery
  Compare the amount of blood loss during the two operations
incidence of surgical complications | One hour to 24 hours after surgery
  delayed hemorrhage, biliary tract injury, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Luhe Hospital affiliated to the Capital Medical University, Beijing, Tongzhou, China

IPD SHARING:
Plan to Share IPD: No